CLINICAL TRIAL: NCT06203548
Title: Monitoring Changes in Hepatic Steatosis During a Lifestyle Intervention Programme in Patients With Non-alcoholic Fatty Liver Disease Using the Novel Continuous Controlled Attenuation Parameter Versus MRI Proton Density Fat Fraction
Brief Title: Monitoring Changes in Hepatic Steatosis Using Continuous Controlled Attenuation Parameter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Vincent WS Wong, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.436
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Intervention Model Description: Lifestyle intervention programme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic dysfunction-associated steatotic liver disease (Other): Adult patients with intrahepatic triglyceride content >=5% by MRI-PDFF
  Interventions: Behavioral: Lifestyle modification programme

INTERVENTIONS:
Behavioral: Lifestyle modification programme — All patients will attend sessions weekly in the first 2 months and monthly in the remaining 4 months. The programme focuses on reducing caloric intake and increasing energy expenditure. At the first visit, the dietitian will perform a complete behavioural assessment including the patient's eating and lifestyle patterns, specific eating-related behaviours, knowledge, concerns and feelings. A target body weight will be set. During follow-up visits, the dietitian will review the patient's dietary pattern and provide recommendations. Each patient will be given an individualised meal plan. The dietary component and portion size are based on recommendations by the American Dietetic. The patients will be taught techniques to cope with at-risk situations such as parties and festival celebrations. In addition, the patients will be encouraged to have a combination of aerobic exercise and resistance training with intensity and frequency following the Physical Activity Guidelines.

SUMMARY:
Background: Non-alcoholic fatty liver disease (NAFLD) affects 30% of the Asian adult population and is emerging as one of the important leading causes of liver cancer and cirrhosis. Although a number of biomarkersmany have been developed for the assessment of liver fat and fibrosis, most existing studies were cross-sectional in nature. The role of these biomarkers for monitoring and response assessment remains elusive. At present, magnetic resonance imaging proton density fat fraction (MRI-PDFF) is considered the gold standard to in quantifying liver fat. The MRI-PDFF response, defined as a ≥30% relative reduction in liver fat fraction, has been shown to correlate with improved hepatic inflammation and fibrosis. However, MRI is limited by cost and availability. The cContinuous controlled attenuation parameter (CAPc) measurement by vibration controlled transient elastography is a new technology to quantify liver fat. It is a point-of-care test and has the potential to replace the MRI-PDFF as a monitoring and response biomarker in routine practice.

Study plan: This prospective cohort study will include 150 patients with NAFLD who will join a 6-month lifestyle modification programme involving dietary intervention and physical training. This will create a cohort of varying degrees of liver fat reduction. Using MRI-PDFF as the reference standard, we will evaluate the accuracy of a changes in CAPc in reflecting the MRI-PDFF response and remission of NAFLD, with all non-invasive tests performed at screening and Month 6. In addition, we will test the hypothesis that the the change in CAPc is superior to the change of in other steatosis tests results (including the original CAP, abdominal ultrasonography and steatosis scores of fatty liver index, hepatic steatosis index, NAFLD liver fat score and NAFLD ridge score) in predicting the MRI-PDFF response. The area under the receiver-operating characteristics curve of the CAPc response in predicting the MRI-PDFF response will be compared with that of the other steatosis tests using the DeLong test.

DETAILED DESCRIPTION:
STUDY DESIGN OVERVIEW In order to evaluate the use of continuous CAP to monitor changes in liver fat over time, we need a cohort of patients with varying degree of liver fat reduction. Therefore, we will enrol MASLD patients in a lifestyle intervention programme. With this design, we will measure original CAP, continuous CAP and MRI-PDFF in all patients at baseline and Month 6. As described in the introduction, MRI-PDFF is an accurate and reliable non-invasive test to quantify liver fat and will serve as the reference standard in this study.

5. CLINIC VISITS AND ASSESSMENTS Clinic visits The patients will attend 4 clinic visits (screening, baseline, month 3 and month 6).

Procedures at the screening visit

* Obtain informed written consent
* Verify conformance with the study inclusion and exclusion criteria
* Record medical history
* Record smoking and alcohol consumption with standard questionnaires
* Physical examination
* Blood tests including complete blood count, prothrombin time, renal function test and liver biochemistry (including alanine aminotransferase [ALT], aspartate aminotransferase [AST] and gamma-glutamyl transpeptidase [GGT]), lipids, plasma glucose and HbA1c.
* Hepatitis B surface antigen and anti-hepatitis C virus antibody
* Vibration-controlled transient elastography examination
* Bedside abdominal ultrasonography. The diagnosis of fatty liver will be based on the presence of bright liver echotexture, deep attenuation of ultrasound signal and blurring of hepatic vasculature.(19)
* Arrange MRI-PDFF examination within 1 week of VCTE examination. The short interval is to avoid significant change in liver fat between the non-invasive measurements of liver fat by original CAP, continuous CAP and MRI-PDFF.

Procedures at the baseline visit

* Verify conformance with the study inclusion and exclusion criteria based on additional laboratory and MRI-PDFF results
* Document new symptoms and adverse events, if any
* Record smoking and alcohol consumption with standard questionnaires
* Document dietary intake over a 1-week period using a locally validated food frequency questionnaire(20)
* Complete the International Physical Activity Questionnaire
* Physical examination including measurement of the patient's body height, body weight, waist circumference, hip circumference and blood pressure
* Body composition measurement
* After overnight fasting for at least 8 hours, blood tests including complete blood count, prothrombin time, renal function test, liver biochemistry including ALT, AST and GGT, plasma glucose, HbA1c, insulin and neuregulin 4.
* and lipid profile including high density lipoprotein (HDL)- and low density lipoprotein (LDL)-cholesterol
* Serum, plasma, and buffy coat samples will be stored for 15 years for future biochemical and genetic studies (optional with separate consent)

Month 3 visit

* Document new symptoms and adverse events, if any
* Record smoking and alcohol consumption with standard questionnaires
* Document dietary intake over a 1-week period using a locally validated food frequency questionnaire(20)
* Complete the International Physical Activity Questionnaire
* Physical examination including measurement of the patient's body height, body weight, waist circumference, hip circumference and blood pressure
* Body composition measurement
* After overnight fasting for at least 8 hours, blood tests including complete blood count, prothrombin time, renal function test, liver biochemistry including ALT, AST and GGT levels, plasma glucose, HbA1c, insulin, neuregulin 4 and lipid profile including HDL- and LDL-cholesterol
* Serum and plasma samples will be stored for 15 years for future biochemical studies (optional with separate consent)
* Vibration-controlled transient elastography examination

Month 6 visit (end of study)

* Document new symptoms and adverse events, if any
* Record smoking and alcohol consumption with standard questionnaires
* Document dietary intake over a 1-week period using a locally validated food frequency questionnaire(20)
* Complete the International Physical Activity Questionnaire
* Physical examination including measurement of the patient's body height, body weight, waist circumference, hip circumference and blood pressure
* Body composition measurement
* After overnight fasting for at least 8 hours, blood tests including complete blood count, prothrombin time, renal function test, liver biochemistry including ALT, AST and GGT levels, plasma glucose, haemoglobin A1c, insulin, neuregulin 4 and lipid profile including HDL- and LDL-cholesterol
* Serum and plasma samples will be stored for 15 years for future biochemical studies (optional with separate consent)
* Bedside abdominal ultrasonography. The diagnosis of fatty liver will be based on the presence of bright liver echotexture, deep attenuation of ultrasound signal and blurring of hepatic vasculature.(19)
* Vibration-controlled transient elastography examination
* Arrange MRI-PDFF examination within 1 week

Lifestyle modification programme In order to produce a patient cohort with various degree of liver fat reduction over time, the patients will participate in a lifestyle modification programme led by dietitians for 6 months. Details of the programme have been described.(6) All patients will attend sessions weekly in the first 2 months and monthly in the remaining 4 months. The programme focuses on reducing caloric intake and increasing energy expenditure. At the first visit, the dietitian will perform a complete behavioural assessment including the patient's eating and lifestyle patterns, specific eating-related behaviours, knowledge, concerns and feelings. A target body weight will be set. During follow-up visits, the dietitian will review the patient's dietary pattern and provide recommendations. Each patient will be given an individualised meal plan. The dietary component and portion size are based on recommendations by the American Dietetic Association with emphasis on fruit and vegetables, moderate-carbohydrate, low-fat, low-glycaemic index and low-calorific products in appropriate portions. The patients will be taught techniques to cope with at-risk situations such as parties and festival celebrations. In addition, the patients will be encouraged to have a combination of aerobic exercise and resistance training with intensity and frequency following the Physical Activity Guidelines.(21)

Vibration controlled transient elastography CAP and liver stiffness will be measured by vibration controlled transient elastography (FibroScan, Echosens, Paris, France) by operators who have performed at least 500 examinations in the past according to the training and instructions by the manufacturer.(22) Our centre is equipped with both the FibroScan 502 Touch and FibroScan 630 Expert machines. The former is used for original CAP measurements, whereas the latter is equipped with the SmartExam software and can be used for continuous CAP measurements. We will choose the M or XL probes according to the machine's automatic probe selection tool.

MRI-PDFF We will perform MRI-PDFF within 1 week from the clinic visit and transient elastography examination. We will use a 3T whole-body scanner (Achieva TX, Philips Healthcare, the Netherlands).(23) We will use the MRI machine that belongs to The Chinese University of Hong Kong. Thus, the study will not affect the service of the hospital. The protocol uses a gradient echo sequence with a low flip angle to minimize T1 bias, and it acquires multiple echoes in which fat and water signals are in or out of phase with respect to each other. After acquiring the data at each echo, an algorithm estimates and corrects T2* effects and calculates the liver fat content by estimating fat and water proton densities. The field of view for the sequences to used will cover the whole abdomen from the xiphoid process to the symphysis pubis to include the whole liver, pancreas, and whole abdominal subcutaneous/visceral adipose tissue. Fatty liver is defined as an intrahepatic triglyceride content of 5% or more. Two operators will analyse the MRI-PDFF results (for liver and pancreatic fat) to ensure a high inter-observer agreement. Additionally, a non-breath-hold acquisition will be performed from the base of the skull to the base of the thoracic cavity for neck and supraclavicular adipose tissue measurements (including brown adipose tissue).

Steatosis scores Based on the clinical and laboratory parameters obtained at baseline and Month 6, we will calculate steatosis scores to determine the presence and resolution of MASLD (Appendix).

Abdominal ultrasonography Abdominal ultrasonography will be performed on the same day as clinical assessment by experienced hepatologists or radiographers who are blinded to all clinical and laboratory data. The examination will be performed using a 5 MHz transducer and a high-resolution B-mode scanner. To ensure consistency across the participating sites, we will use the Hamaguchi system to score the liver for (1) bright liver and hepatorenal echo contrast (0-3 points), (2) deep attenuation (0-2 points), and (3) vessel blurring (0-1 point).(19) A score of ≥2 has 92% sensitivity and 100% specificity for the diagnosis of MASLD.

For exploratory purpose, attenuation imaging (ATI) during ultrasonography will be performed in around half of the subjects (n=75). An Aplio i800, Canon medical systems, Tochigi, Japan ultrasound machine will be used. Using a 1 to 8MHz convex transducer (i8CX1), the liver parenchyma will be first evaluated on B-mode to ensure that the fan shaped sampling box is placed in a homogenous region, thereafter the ATI mode will be activated. All images will be obtained in the supine position and in the intercostal planes with the transducer perpendicular to the skin. An approximately 4 x 8cm sampling box will be positioned randomly in the liver (including the left lobe), 2 cm below the capsule during several seconds of breath-holding. Non-homogeneous areas such as large vessels and cystic structures are automatically excluded from the ATI map using a system inherent structure removal filter. Thus, homogenous ATI colour maps will be acquired as much as possible. By careful avoidance of large vessels and areas of reverberation artifacts, a 2 x 4cm region of interest for measurement will be set within the sampling box of ATI and placed in the middle portion of the sampling box to reduce the intra-observer variability. Attenuation Coefficient with R2 ≥ 0.92 will be regarded as valid measurement. ATI examinations will be performed in five valid Attenuation Coefficient (dB/cm/MHz) measurements, of which the median value of the measurements will be used for analysis. The estimated scan time is 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Intrahepatic triglyceride content by MRI-PDFF ≥5%
* At least one metabolic risk factor out of (1) body-mass index ≥23 kg/m2, (2) waist circumference ≥90 cm in men and ≥80 cm in women, (3) fasting plasma glucose ≥5.6 mmol/L, 2-hour post-load glucose ≥7.8 mmol/L, haemoglobin A1c (HbA1c) ≥5.7%, known diabetes or on treatment for type 2 diabetes, (4) blood pressure ≥130/85 mmHg or on treatment for hypertension, (5) plasma triglycerides ≥1.7 mmol/L or on treatment for dyslipidaemia, and (6) plasma high-density lipoprotein-cholesterol ≤1.0 mmol/L in men and ≤1.3 mmol/L in women or on treatment for dyslipidaemia
* Provide informed written consent

Exclusion Criteria:

* Positive hepatitis B surface antigen or anti-hepatitis C virus antibody, or history or evidence of other liver diseases
* Alcohol consumption >30 g per day in men or >20 g per day in women
* Liver decompensation, as evidenced by total bilirubin >50 µmol/L (except in patients with documented Gilbert's syndrome), platelet count <100 x 109/L, prothrombin time >1.3 times the upper limit of normal, albumin <35 g/L, or history or presence of ascites, varices or hepatic encephalopathy
* Contraindications to MRI examination such as claustrophobia or the presence of metallic implants
* History or presence of hepatocellular carcinoma
* History of other malignancies, unless in complete remission for more than 5 years
* History of liver transplantation or liver resection
* Significant co-morbidities that will likely limit a patient's participation in lifestyle intervention or attendance of study follow-ups

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
MRI-PDFF response | 6 months
  >30% relative reduction in MRI-PDFF

SECONDARY OUTCOMES:
Remission of MASLD | 6 months
  Liver fat fraction by MRI-PDFF <5%

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No